CLINICAL TRIAL: NCT02302950
Title: A Retrospective Analysis of Raltegravir Use in Minority HIV Infected Women in Houston, Texas
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tanvir K. Bell, MD, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0559
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection
Keywords: HIV infection; raltegravir use; women
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women that picked up raltegravir 2013: minority women that picked up raltegravir at Thomas street Health Center 2013
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — HIV therapy component
  Other Names: issentress

SUMMARY:
Raltegravir is the first marketed strand-transfer inhibitor of HIV-1 that was FDA approved in 2007. It is currently one of the preferred treatment regimens for HIV by the Department of Health and Human Services. It has become a widely used antiretroviral therapy option for HIV infected patients. It provides good tolerability and a favorable lipid profile for patients when compared to some other antiretroviral treatment options. Little data is reported about efficacy in a minority patient population. Moreover, data in an indigent minority population in the United States has not been aggregated before. Therefore this study will investigate the efficacy of raltegravir in minority women residing in Houston, TX who are HIV infected.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected women who picked up raltegravir in the year 2013 at Thomas Street Health Center.
2. Minority women -Black/African American, Hispanic/Latino

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected minority women at Thomas Street Health Center that picked up raltegravir in 2013
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of raltegravir in study participants by measuring CD4 count and viral load | 24 weeks of therapy

SECONDARY OUTCOMES:
Capture data on concomitant conditions that may have led to participants switching to raltegravir from medical records (eg. Diabetes mellitus) | 24 weeks of therapy
Assess tolerability of raltegravir by capturing symptoms | 24 weeks of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Street Clinic, Houston, Texas, United States